CLINICAL TRIAL: NCT04900207
Title: Placental Volume, Flow, and Vascularity Study
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00009133
Record Dates: First submitted 2021-04-26; First posted 2021-05-25 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed Group: Participants will be enrolled in the study at the time of their first-trimester screen (10w3d-13w6d weeks of gestation) to the time of their delivery. Collection of first-trimester 3D-volume ultrasound imaging to measure the placental volume, blood flow, and vascularity and maternal serum markers will occur over a 6-12 months period. Collection of descriptive and pregnancy outcome information will be obtained from the electronic medical records will continue through their pregnancy episode (typical 9 months).

SUMMARY:
The purpose of this preliminary study is to implement an automated and standardized computer-based method that accurately measures placental volume, blood flow, and vascularity. This will be accomplished by using the digital data obtained at the time of a first-trimester 3D image volume. This information will then be used to further investigate whether placental volume, blood flow, and vascularity can be used to predict the risk of preeclampsia in conjunction with maternal history and serum blood markers obtained at the time of their ultrasound.

DETAILED DESCRIPTION:
Preeclampsia is defined as a multi-system disorder typically characterized by hypertension, proteinuria, and/or end organ damage. Preeclampsia can develop rapidly at any time after 20 weeks gestation and into the postpartum period and can at times lead to systemic complications and even death. Preeclampsia continues to be a leading cause of maternal morbidity and mortality secondary to the development of hypertensive disorders, systemic inflammatory changes affecting the endothelium, and hemorrhagic complications. It also contributes indirectly to neonatal morbidity and mortality by leading to premature delivery. Our current ability to screen patients for the risk of developing preeclampsia relies on clinical factors as recommended by ACOG and the USPHS. At this time, if a patient is deemed high risk, our only intervention for prevention of preeclampsia is to prescribe low-dose aspirin. Being able to identify the population at higher risk for preeclampsia would allow for implementation of new management options among these persons. The purpose of this preliminary study is to implement an automated and standardized computer-based method that accurately measures placental volume, blood flow, and vascularity. This will be accomplished by using the digital data obtained at the time of a first-trimester 3D image volume. This information will then be used to further investigate whether placental volume, blood flow, and vascularity can be used to predict the risk of preeclampsia in conjunction with maternal history and serum blood markers obtained at the time of their ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Qualify for a first-trimester screen at the time of enrollment. Criteria for the screen include pregnancy with gestational age between 10 weeks 3 days and 13 weeks 6 days of gestation as well as a crown-rump length between 40 and 84 mm.
* Complete a first-trimester ultrasound at the qualifying M Health Fairview Maternal Fetal Medicine Clinics, which include University Riverside, Ridges, South Dale, and Health East sites
* Provide a blood sample for either completion of the first-trimester screen and/or for the completion of the research study

Exclusion Criteria:

* Multi-fetal gestation or pregnancy with major fetal congenital anomalies and/or known fetal aneuploidy
* Unwilling to complete a first-trimester ultrasound and/or unwilling to provide a serum sample

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants are pregnant adults in the first trimester of gestation who are receiving an ultrasound at one of the qualifying study sites.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Predictive Value of Model for the Development of Preeclampsia | up to 12 months
  The primary measure for this study will be the positive predictive value of the model for the development of preeclampsia. Outcome is reported as the percent of correct predictions made by the model.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Contag, MD, Principal Investigator — University of Minnesota Medical School Department of Obstetrics, Gynecology, & Women's Health
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No